CLINICAL TRIAL: NCT04385797
Title: Cognitive Outcomes During COVID-19 confiNemeNt in Elderly and Their Caregivers Using Technologies for DEMentia
Acronym: CONNECTDEM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Other Study IDs: CONNECT DEM
Record Dates: First submitted 2020-05-07; First posted 2020-05-13 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-04

CONDITIONS: Mild Cognitive Impairment; Dementia
Keywords: COVID-19; Social Isolation; Informal caregivers; Cognition; Facilities and Services Utilization; Technologies; ICTs; Telehealth
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; COVID-19; Social Isolation | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dyads: Community-dwelling older adults with mild cognitive impairment or mild dementia and their caregivers
  Interventions: Other: Telephone interview

INTERVENTIONS:
Other: Telephone interview — Sociodemographic data. Clinical data. PMCI/MD quality of life, cognition, depression, technophilia and perceived stress and caregiver quality of life and burden assessments.

SUMMARY:
Coronavirus disease 2019 has forced worldwide the implementation of unprecedented restrictions to control its rapid spread and mitigate its impact. The Spanish government has enforced social distancing, quarantine and home confinement. This restriction of daily life activities and separation from loved ones may lead to social isolation and loneliness with health-related consequences in community-dwelling older adults with mild cognitive impairment or mild dementia and their caregivers. Additionally, an inadequate access to healthcare and social support services may aggravate chronic conditions. Technology home-based interventions emerge for combating social isolation and loneliness preventing the risk of viral exposure.

The aim of this multicentre cohort study is to explore, analyze and determine the impact of social isolation on: 1) cognition, quality of life, mood, technophilia and perceived stress of community-dwelling older adults with mild cognitive impairment or mild dementia, and on caregiver burden; 2) health and social care services access and utilization, and 3) cognitive, social and entertainment use of ICTs.

This study will be conducted in two Spanish regions Andalucía (Málaga) and Cataluña (Tarrasa). In total 200 dyads, consisting of a person with mild cognitive impairment or mild dementia (PMCI/MD) and their informal caregiver will be contacted by telephone. Potential respondents will be participants of the SMART 4 MD (N=100) and TV-AssistDem (N=100) clinical trials.

The change in means in the variables will be analyzed comparing baseline results in the previous studies with those during and after confinement using the ANOVA test of repeated measures or the non-parametric Friedman test if appropriate. The performance of a multivariate analysis of variance (ANCOVA) to introduce possible covariates will also be contemplated. A 95% confidence level will be used.

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19) has forced worldwide government authorities to implement unprecedented restrictions to control its rapid spread and mitigate its impact. In response to the outbreak, Spain declared by royal decree (463/2020) a national emergency, with the exceptional measure of a Nationwide lockdown enforcing social distancing, quarantine of those exposed to the disease and home confinement of those who remain healthy allowing only essential outings. This home-confinement by restriction of movement of daily life activities and social distancing from loved ones may be a challenging and unpleasant experience for those who undergo it, experiencing social isolation and loneliness with health-related consequences. Vulnerable populations at higher risk are fragile community-dwelling older adults whose chronic conditions may be aggravated by the consequences of the confinement and in particular, people with mild cognitive impairment or mild dementia.

QUALITY ASSURANCE PLAN. Researchers will report and review the process during the trial covering participant enrolment, consent, follow-up, policies to protect participants, including reporting of harm and completeness, accuracy, and timelines of data collection.

STANDARD OPERATING PROCEDURES. Participants will be interviewed by telephone. Potential respondents will be participants of the SMART 4 MD (NCT03325699) and TV-AssistDem (NCT03653234) clinical trials, which all aim to assess the effects of ICTs to support dementia: using a tablet-based health application, an intelligent system and a TV-based assistive integrated service, respectively.

Baseline assessments prior to the COVID-19 confinement (T0) of cognition, quality of life, depression, and technophilia of the PMCI/MD and caregiver burden will be compared with assessments carried out during the confinement measures (T1) and after the termination of the measures (T2). Additionally, perceived stress regarding the confinement situation will be measured at T1 and T2.

Participants will not receive financial reimbursement for taking part in this trial.

DATA DICTIONARY. All variables collected in this study are listed and described in an electronic Case Report Form (CRF), with associated guidelines, to ensure consistency in all gathered data. The following data will be collected in this trial:

Mini-Mental State Examination (MMSE) Quality of Life-Alzheimer's Disease Scale (QoL-AD Scale) European Quality of Life 5 Dimensions 3 Levels (EuroQoL-5D-3L) Geriatric Depression Scale (GDS) Instrument for Measuring Older People's Attitudes Toward Technology (TechPH) Perceived Stress Scale (PSS) Zarit Burden Interview (ZBI-12)

Other data: Sociodemographical data. Medical history - PMCI/MD only. Health perception-management: Change of living arrangements due to lockdown, presence of COVID-19 symptoms in PMCI/MD and/or relatives, access to COVID-19 information, devices used (SmartPhone, Tablet, Computer, Smart-TV, other), understanding of the information and contact with healthcare and social resources to manage the situation. Ability to manage illnesses, medication, changes and/or cancellations of previous medical appointments, renewal of prescriptions and provision of supports for the purchase of medication and food. Coping-stress tolerance: Mental health and well-being self-perceived mood. Sleep-rest : Alterations in usual sleep patterns and use of additional medication. Leisure activities: including preferred physical, intellectual, recreational and social activities. Social support: social connectedness (telephone call, video call, texting...), devices used (SmartPhone, Tablet, Computer, Smart-TV, other)

STATISTICS ANALYSIS PLAN. The flow of participants will be shown schematically with counts and percentages in a CONSORT diagram. All variables collected will be summarized at baseline and at follow-up. Statistics considered for presentation for continuous measures in summary tables will be the mean, minima and maxima, and standard deviation, and if the criteria of normality are not met, the median and the first and third quartiles. Categorical variables will be summarized using counts and percentages. The change in means in the study variables will be analyzed with respect to the results during the previous studies (SMART 4 MD and TV-AssistDem) with those currently collected using the ANOVA test of repeated measures or the non-parametric Friedman test if appropriate. The performance of a multivariate analysis of variance (ANCOVA) to introduce possible covariates will also be contemplated. A 95% confidence level will be used for all comparisons. The R version 3.6.1 program will be used. for all statistical analysis.

PLAN FOR MISSING DATA. Each researcher is responsible for ensuring that any missing data will be reported as missing in the study database. Procedures can sometimes be considered when using statistical methods that fail in the presence of any missing values, or when in the case of multiple-predictor statistical models all the data for an individual would be omitted because of a missing value in one of the predictors.

METHODS TO ENSURE VALIDITY AND QUALITY OF DATA. Accurate and reliable data collection will be assured by verification and cross-check of the CRF. Discrepancies and queries will be generated accordingly in the CRF for online resolution by the researcher. In addition, the CRF data will be reviewed on an ongoing basis for scientific plausibility.

ELIGIBILITY:
Inclusion Criteria:

* Having participated in the SMART 4 MD, TV-AssistDem and INFINITy clinical trials

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community-dwelling older adults with mild cognitive impairment or mild dementia
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Change on cognitive function in people with mild cognitive impairment or mild dementia prior to, during and after confinement. | Through study completion, an average of 6 months
  The Mini-Mental State Examination (MMSE) (23) will be used to assess the cognitive function of the PMCI/MD. The most common cutoff scores for cognitive impairment and dementia are ranging 23 to 27 over 30. As telephone call interviewing will be the safest means to communicate with the PMCI/MD during and after the COVID-19 pandemic the 22 items telephone version of the MMSE will be used (24). All points of the MMSE can be covered in the telephone version except the last section assessing language and motor skills. In the phone version, we will ask the subject to repeat a phrase and name one item (For example: "Tell me, what is the name of the object you are using to talk to me?"). However, a second item will be not be named, nor will be the person be asked to follow a three-stage command, read and obey a sentence, write a sentence, or copy an intersecting pentagon as in the original version.

SECONDARY OUTCOMES:
Change on quality of life in Alzheimer´s Disease in people with mild cognitive impairment or mild dementia prior to, during and after confinement. | Through study completion, an average of 6 months
  The Quality of Life-Alzheimer's Disease Scale (QoL-AD) (19-22) is an instrument specifically designed to measure QoL in PMCI/MD from the perspective of both the patient and the informal caregiver. It is a 13-item measure, which includes assessments of the person´s relationships with friends and family, financial situation, physical condition, mood, memory, and an overall assessment of life quality. Response are 4-point multiple choice options (1 = poor, 2= fair, 3= good, 4 = excellent). Scale scores range from 13 to 52, with higher scores indicating greater quality of life.
  When cognitive function may be compromised, informal caregivers will complete the QoL-AD, on behalf of the PMCI/MD.
Change on quality of life in people with mild cognitive impairment or mild dementia prior to, during and after confinement. | Through study completion, an average of 6 months
  The European Quality of Life 5 Dimensions 3 Levels (EuroQoL-5D-3L) is a standardized generic instrument consisting of a descriptive system and a visual analogue scale (VAS).
  The descriptive system comprises 5 dimensions covering mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, moderate problems and extreme problems. A 1-digit number expresses the level selected for that dimension. The digits can be combined into a 5-digit number that describes the patient's health state.
  The VAS records the patient's self-rated health on a vertical scale, where the endpoints are 100 = 'The best health you can imagine' and 0 = 'The worst health you can imagine'.
  EuroQoL-5D-3L has been shown to correlate well with QoL-AD, indicating that using both measures side-by-side is compatible.
Change on mood in people with mild cognitive impairment or mild dementia prior to, during and after confinement. | Through study completion, an average of 6 months
  The Short Form of the Geriatric Depression Scale (GDS) (25) will be used to assess mood. Of the 15 items, 10 indicate depression when answered positively, while the rest (1, 5, 7, 11, 13) when answered negatively. Scores of 0-4 are considered normal, 5-8 indicate mild depression, 9-11 moderate depression, and 12-15 severe depression.
Change on technophilia in people with mild cognitive impairment or mild dementia prior to, during and after confinement. | Through study completion, an average of 6 months
  The Instrument for Measuring Older People's Attitudes Toward Technology (TechPH) measures older people's attitudes and enthusiasm for health technology (26). This instrument refers to technophilia as a person's enthusiasm for and positive feelings toward their technology use and absence of the fears and doubts some older people could have about their ability to manage using new technology. The six items of the instrument measure two factors of technophilia: 3 items concerning techEnthusiasm and 3 items techAnxiety. Response are constructed with a five-point Likert scale questionnaire, ranging from 1 (fully disagree) to 5 (fully agree).
Change on perceived stress in people with mild cognitive impairment or mild dementia during and after confinement. | Through study completion, an average of 6 months
  The Perceived Stress Scale (PSS) measures the degree to which situations in one's life are appraised as stressful. The scale has 10 questions regarding feelings and thoughts during the last month and are rated according to frecuency 0 = Never 1 = Almost Never 2 = Sometimes 3 = Fairly Often 4 = Very Often. PSS scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the four positively stated items (items 4, 5, 7, & 8) and then summing across all scale items
Change on caregiver burden prior to, during and after confinement. | Through study completion, an average of 6 months
  The Zarit Burden Interview (ZBI-12) is a 12-item scale with each answer chosen from a 5-point Likert scale (Nearly always=4, Quite frequently=3, Sometimes=2, Rarely=1, Never=0). It is a shortened version of the original scale, was developed specifically for informal caregivers of PMCI/MD and covers issues such as caregiver stress and the degree to which caring is affecting their health and social life. Total score range 0 to 48 (0-10= no to mild burden, 10-20= mild to moderate burden >20= high burden).
Change on healthcare and social support services access prior to, during and after confinement. | Through study completion, an average of 6 months
  The Client Service Receipt Inventory (CSRI) (32,33) scale will be used to evaluate the service utilization. This scale is an internationally used method for gathering data on service utilization and other domains relevant for economic analysis of mental health care. It has five sections: background client information, accommodation and living situation, employment history, earnings and benefits, a record of services usually used and information about informal caregiver support. The sections assessed will be consultations, admissions and visits, grouped into subsections according to hospital, specialist, primary or home care. Treatment related to hospital admissions or illness exacerbation will also be assessed. It´s adaptability ensures it is compatible with the research aims, context, participants' likely circumstances, and the quantity and precision of information required.
Change from health, cognitive, social, informative and entertainment related uses of ICT during and after confinement. | Through study completion, an average of 6 months
  Use of ICTs (SmartPhone, Tablet, Computer, Smart-TV, or other) to contact healthcare and social support services, to stimulate cognition, to facilitate social connectedness (telephone call, video call, texting...), to access COVID-19 information and to enable entertainment.

CONTACTS AND LOCATIONS:
Overall Officials: Fermín Mayoral-Cleries, Principal Investigator — Instituto de Investigación Biomédica de Malaga (IBIMA)
Locations (1):
- Instituto de Investigacion Biomedica de Malaga-IBIMA, Málaga, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sohrabi C, Alsafi Z, O'Neill N, Khan M, Kerwan A, Al-Jabir A, Iosifidis C, Agha R. World Health Organization declares global emergency: A review of the 2019 novel coronavirus (COVID-19). Int J Surg. 2020 Apr;76:71-76. doi: 10.1016/j.ijsu.2020.02.034. Epub 2020 Feb 26. PMID 32112977
- [Background] Legido-Quigley H, Mateos-Garcia JT, Campos VR, Gea-Sanchez M, Muntaner C, McKee M. The resilience of the Spanish health system against the COVID-19 pandemic. Lancet Public Health. 2020 May;5(5):e251-e252. doi: 10.1016/S2468-2667(20)30060-8. Epub 2020 Mar 18. No abstract available. PMID 32199083
- [Background] Brooks SK, Webster RK, Smith LE, Woodland L, Wessely S, Greenberg N, Rubin GJ. The psychological impact of quarantine and how to reduce it: rapid review of the evidence. Lancet. 2020 Mar 14;395(10227):912-920. doi: 10.1016/S0140-6736(20)30460-8. Epub 2020 Feb 26. PMID 32112714
- [Background] World Health Organization. Mental Health and Psychosocial Considerations During COVID-19 Outbreak. World Heal Organ 2020;(January):1-6.
- [Background] Gomez-Gallego M, Gomez-Amor J, Gomez-Garcia J. [Validation of the Spanish version of the QoL-AD Scale in alzheimer disease patients, their carers, and health professionals]. Neurologia. 2012 Jan;27(1):4-10. doi: 10.1016/j.nrl.2011.03.006. Epub 2011 May 12. Spanish. PMID 21570161
- [Background] Garcia-Gordillo MA, Adsuar JC, Olivares PR. Normative values of EQ-5D-5L: in a Spanish representative population sample from Spanish Health Survey, 2011. Qual Life Res. 2016 May;25(5):1313-21. doi: 10.1007/s11136-015-1164-7. Epub 2015 Oct 19. PMID 26482825
- [Background] Anderberg P, Eivazzadeh S, Berglund JS. A Novel Instrument for Measuring Older People's Attitudes Toward Technology (TechPH): Development and Validation. J Med Internet Res. 2019 May 23;21(5):e13951. doi: 10.2196/13951. PMID 31124467
- [Background] Remor E. Psychometric properties of a European Spanish version of the Perceived Stress Scale (PSS). Span J Psychol. 2006 May;9(1):86-93. doi: 10.1017/s1138741600006004. PMID 16673626
- [Background] Bedard M, Molloy DW, Squire L, Dubois S, Lever JA, O'Donnell M. The Zarit Burden Interview: a new short version and screening version. Gerontologist. 2001 Oct;41(5):652-7. doi: 10.1093/geront/41.5.652. PMID 11574710
- [Background] Fernandez-San Martin M, Andrade-Rosa C, Molina JD, Munoz PE, Carretero B, Rodriguez M, Silva A. Validation of the Spanish version of the geriatric depression scale (GDS) in primary care. Int J Geriatr Psychiatry. 2002 Mar;17(3):279-87. doi: 10.1002/gps.588. PMID 11921157
- [Background] Tsoi KKF, Chan JYC, Hirai HW, Wong A, Mok VCT, Lam LCW, Kwok TCY, Wong SYS. Recall Tests Are Effective to Detect Mild Cognitive Impairment: A Systematic Review and Meta-analysis of 108 Diagnostic Studies. J Am Med Dir Assoc. 2017 Sep 1;18(9):807.e17-807.e29. doi: 10.1016/j.jamda.2017.05.016. Epub 2017 Jul 25. PMID 28754516
- [Derived] Dura-Perez E, Goodman-Casanova JM, Vega-Nunez A, Guerrero-Pertinez G, Varela-Moreno E, Garolera M, Quintana M, Cuesta-Vargas AI, Barnestein-Fonseca P, Gomez Sanchez-Lafuente C, Mayoral-Cleries F, Guzman-Parra J. The Impact of COVID-19 Confinement on Cognition and Mental Health and Technology Use Among Socially Vulnerable Older People: Retrospective Cohort Study. J Med Internet Res. 2022 Feb 22;24(2):e30598. doi: 10.2196/30598. PMID 35049505
- [Derived] Goodman-Casanova JM, Dura-Perez E, Guerrero-Pertinez G, Barnestein-Fonseca P, Guzman-Parra J, Vega-Nunez A, Varela-Moreno E, Cuesta-Vargas A, Mayoral-Cleries F. Cognitive Outcomes During COVID-19 Confinement Among Older People and Their Caregivers Using Technologies for Dementia: Protocol for an Observational Cohort Study. JMIR Res Protoc. 2021 May 18;10(5):e26431. doi: 10.2196/26431. PMID 33909588